CLINICAL TRIAL: NCT01258543
Title: Osteopathic Evaluation on Patients With Non-specific Back Pain: An Observational Inter-examiner Reliability Study
Brief Title: Osteopathic Evaluation on Patients With Non-specific Back Pain: An Inter-examiner Reliability Study
Status: Completed | Type: Observational
Sponsor: Kirnan, Jaime (Individual)
Responsible Party: Jaime Kirnan, Unaffiliated
Other Study IDs: JAK-OST-1
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Inter-examiner Reliability; Location and Nature of Restriction or Lesion; Non-specific Back Pain
Keywords: Global osteopathic evaluation; Non-specific back pain; Inter-examiner reliability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-specific back pain
  Interventions: Other: General Osteopathic Evaluation

INTERVENTIONS:
Other: General Osteopathic Evaluation — 2 general osteopathic evaluations of approximately 1 hour in duration done consecutively on the same day with a 15 minute break between evaluations

SUMMARY:
The purpose of this study is to determine whether two osteopathic evaluators with less than 5 years experience will be able to determine the same location and nature of the primary lesion(s) or restriction(s)in patients with chronic non-specific back pain using a global osteopathic evaluation approach.

DETAILED DESCRIPTION:
Back pain is one of the leading causes of consultation for rehabilitation. Establishing a diagnosis in the initial patient assessment is essential to choosing a specific treatment plan for that patient, regardless of the type of therapy the patient chooses to pursue. Evidence based medicine is the current gold standard for most manual-therapy professions, and there has been a great deal of research performed in an attempt to give credibility to the one tool that all manual therapy professions share in common: palpation. Few studies have been able to demonstrate an acceptable rate of inter-examiner reliability for palpation. This study will combine a global testing regime, consensus training for evaluators, and access to history of injury with symptomatic subjects to verify the inter-examiner reliability of an osteopathic evaluation on patients with chronic, non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-60
* Must have a history of non-specific back pain (not due to any known pathology eg. disc herniation or disc degenerative disease) that is currently not irritated and has not been, in the past 8 weeks
* Must be available for 3 consecutive hour

Exclusion Criteria:

* Patients with a known cause for their back pain
* Patients who have had a flare up of symptoms within the last 8 weeks
* Patients who are currently undergoing any rehabilitation or who have received manual treatment in the last 8 weeks.
* Patients who are taking daily medications for pain
* Pregnant women
* Major medical conditions: fractures, degenerative arthritis, inflammatory disorders, ankylosing spondylitis, multiple sclerosis, cancer, paralysis stroke or recent concussion history
* Any other conditions that would prevent the participant from completing the evaluation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Inter-examiner reliability | Day 1
  Inter-examiner reliability between two evaluators for nature and location of primary restriction(s), lesion(s) found during a global osteopathic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: René Pelletier, MSc., D.O, Study Director; Sabrina Silla, BSc., PT, DO, Study Director; Jaime Kirnan, BSc., CAT(c), Principal Investigator
Locations (1):
- Concordia Physio Sport, Brossard, Quebec, Canada

REFERENCES:
- [Background] Beal MC, Patriquin DA. Interexaminer agreement on palpatory diagnosis and patient self-assessment of disability: a pilot study. J Am Osteopath Assoc. 1995 Feb;95(2):97-100, 103-6. PMID 7890559
- [Background] Bertilson BC, Grunnesjo M, Strender LE. Reliability of clinical tests in the assessment of patients with neck/shoulder problems-impact of history. Spine (Phila Pa 1976). 2003 Oct 1;28(19):2222-31. doi: 10.1097/01.BRS.0000089685.55629.2E. PMID 14520035
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Christensen HW, Vach W, Vach K, Manniche C, Haghfelt T, Hartvigsen L, Hoilund-Carlsen PF. Palpation of the upper thoracic spine: an observer reliability study. J Manipulative Physiol Ther. 2002 Jun;25(5):285-92. doi: 10.1067/mmt.2002.124424. PMID 12072848
- [Background] Cleland JA, Childs JD, Fritz JM, Whitman JM. Interrater reliability of the history and physical examination in patients with mechanical neck pain. Arch Phys Med Rehabil. 2006 Oct;87(10):1388-95. doi: 10.1016/j.apmr.2006.06.011. PMID 17023251
- [Background] Comeaux, Z., Eland, D., Chila, A., Pheley, A., & Tate, M. (2001). Measurement challenges in physical diagnosis: refining inter-rater palpation, perception and communication. Journal of Bodywork and Movement Therapies; 5(4): 245-253
- [Background] Degenhardt BF, Snider KT, Snider EJ, Johnson JC. Interobserver reliability of osteopathic palpatory diagnostic tests of the lumbar spine: improvements from consensus training. J Am Osteopath Assoc. 2005 Oct;105(10):465-73. PMID 16314679
- [Background] French SD, Green S, Forbes A. Reliability of chiropractic methods commonly used to detect manipulable lesions in patients with chronic low-back pain. J Manipulative Physiol Ther. 2000 May;23(4):231-8. doi: 10.1067/mmt.2000.106101. PMID 10820295
- [Background] Fritz JM, Delitto A, Vignovic M, Busse RG. Interrater reliability of judgments of the centralization phenomenon and status change during movement testing in patients with low back pain. Arch Phys Med Rehabil. 2000 Jan;81(1):57-61. doi: 10.1016/s0003-9993(00)90222-3. PMID 10638877
- [Background] Freyer, G., McPherson, H. C., & O'Keefe, P. (2005). The effect of training on the inter-examiner and intra-examiner reliability of the seated flexion test and assessment of pelvic anatomical landmarks with palpation. International Journal of Osteopathic Medicine; 8: 131-138.
- [Background] Ghoukassian, M., Nicholls, B., & McLaughlin, P. (2001). Inter-examiner reliability of the Johnson and Friedman percussion scan of the thoracic spine. Journal of Osteopathic Medicine; 4(1): 15-20
- [Background] Haas M. Interexaminer reliability for multiple diagnostic test regimens. J Manipulative Physiol Ther. 1991 Feb;14(2):95-103. PMID 2019826
- [Background] Haas M. Statistical methodology for reliability studies. J Manipulative Physiol Ther. 1991 Feb;14(2):119-32. PMID 2019821
- [Background] Haas M. The reliability of reliability. J Manipulative Physiol Ther. 1991 Mar-Apr;14(3):199-208. PMID 2045731
- [Background] Hall H, McIntosh G, Boyle C. Effectiveness of a low back pain classification system. Spine J. 2009 Aug;9(8):648-57. doi: 10.1016/j.spinee.2009.04.017. Epub 2009 Jun 4. PMID 19501026
- [Background] Hestbaek L, Leboeuf-Yde C. Are chiropractic tests for the lumbo-pelvic spine reliable and valid? A systematic critical literature review. J Manipulative Physiol Ther. 2000 May;23(4):258-75. doi: 10.1067/mmt.2000.106097. PMID 10820299
- [Background] Hicks GE, Fritz JM, Delitto A, Mishock J. Interrater reliability of clinical examination measures for identification of lumbar segmental instability. Arch Phys Med Rehabil. 2003 Dec;84(12):1858-64. doi: 10.1016/s0003-9993(03)00365-4. PMID 14669195
- [Background] Horneij E, Hemborg B, Johnsson B, Ekdahl C. Clinical tests on impairment level related to low back pain: a study of test reliability. J Rehabil Med. 2002 Jul;34(4):176-82. doi: 10.1080/16501970213235. PMID 12201613
- [Background] Huijbregts, P. A. (2002). Spinal motion palpation: a review of reliability studies. Manipulative and Physiological Therapeutics; 10(1): 24-39
- [Background] Jull G, Zito G, Trott P, Potter H, Shirley D. Inter-examiner reliability to detect painful upper cervical joint dysfunction. Aust J Physiother. 1997;43(2):125-129. doi: 10.1016/s0004-9514(14)60406-2. PMID 11676679
- [Background] Keating JC Jr, Bergmann TF, Jacobs GE, Finer BA, Larson K. Interexaminer reliability of eight evaluative dimensions of lumbar segmental abnormality. J Manipulative Physiol Ther. 1990 Oct;13(8):463-70. PMID 2146357
- [Background] Kokmeyer DJ, Van der Wurff P, Aufdemkampe G, Fickenscher TC. The reliability of multitest regimens with sacroiliac pain provocation tests. J Manipulative Physiol Ther. 2002 Jan;25(1):42-8. doi: 10.1067/mmt.2002.120418. PMID 11898017
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Laslett M, Williams M. The reliability of selected pain provocation tests for sacroiliac joint pathology. Spine (Phila Pa 1976). 1994 Jun 1;19(11):1243-9. doi: 10.1097/00007632-199405310-00009. PMID 8073316
- [Background] Leboeuf-Yde C, Kyvik KO. Is it possible to differentiate people with or without low-back pain on the basis of test of lumbopelvic dysfunction? J Manipulative Physiol Ther. 2000 Mar-Apr;23(3):160-7. doi: 10.1016/s0161-4754(00)90245-8. PMID 10771500
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Maher C, Adams R. Reliability of pain and stiffness assessments in clinical manual lumbar spine examination. Phys Ther. 1994 Sep;74(9):801-9; discussion 809-11. doi: 10.1093/ptj/74.9.801. PMID 8066107
- [Background] Meijne W, van Neerbos K, Aufdemkampe G, van der Wurff P. Intraexaminer and interexaminer reliability of the Gillet test. J Manipulative Physiol Ther. 1999 Jan;22(1):4-9. doi: 10.1016/s0161-4754(99)70098-9. PMID 10029942
- [Background] Mior SA, McGregor M, Schut B. The role of experience in clinical accuracy. J Manipulative Physiol Ther. 1990 Feb;13(2):68-71. PMID 2307923
- [Background] Murphy DR, Hurwitz EL, Nelson CF. A diagnosis-based clinical decision rule for spinal pain part 2: review of the literature. Chiropr Osteopat. 2008 Aug 11;16:7. doi: 10.1186/1746-1340-16-7. PMID 18694490
- [Background] Perreault N, Brisson C, Dionne CE, Montreuil S, Punnett L. Agreement between a self-administered questionnaire on musculoskeletal disorders of the neck-shoulder region and a physical examination. BMC Musculoskelet Disord. 2008 Mar 17;9:34. doi: 10.1186/1471-2474-9-34. PMID 18366656
- [Background] Pool JJ, Hoving JL, de Vet HC, van Mameren H, Bouter LM. The interexaminer reproducibility of physical examination of the cervical spine. J Manipulative Physiol Ther. 2004 Feb;27(2):84-90. doi: 10.1016/j.jmpt.2003.12.002. PMID 14970808
- [Background] Robinson HS, Brox JI, Robinson R, Bjelland E, Solem S, Telje T. The reliability of selected motion- and pain provocation tests for the sacroiliac joint. Man Ther. 2007 Feb;12(1):72-9. doi: 10.1016/j.math.2005.09.004. Epub 2006 Jul 12. PMID 16843031
- [Background] Schneider M, Erhard R, Brach J, Tellin W, Imbarlina F, Delitto A. Spinal palpation for lumbar segmental mobility and pain provocation: an interexaminer reliability study. J Manipulative Physiol Ther. 2008 Jul-Aug;31(6):465-73. doi: 10.1016/j.jmpt.2008.06.004. PMID 18722203
- [Background] Seffinger MA, Najm WI, Mishra SI, Adams A, Dickerson VM, Murphy LS, Reinsch S. Reliability of spinal palpation for diagnosis of back and neck pain: a systematic review of the literature. Spine (Phila Pa 1976). 2004 Oct 1;29(19):E413-25. doi: 10.1097/01.brs.0000141178.98157.8e. PMID 15454722
- [Background] Seffinger, M., Adams, A., Najm, W., Dickerson, V., Mishra, S. I., Reinsch, S., & Murphy, L. (2003). Spinal palpatory diagnostic procedures utilized by practitioners of spinal manipulation: annotated bibliography of content validity and reliability studies. Journal of the Canadian Chiropractic Association; 47(2): 93-109
- [Background] Smedmark V, Wallin M, Arvidsson I. Inter-examiner reliability in assessing passive intervertebral motion of the cervical spine. Man Ther. 2000 May;5(2):97-101. doi: 10.1054/math.2000.0234. PMID 10903585
- [Background] Stochkendahl MJ, Christensen HW, Hartvigsen J, Vach W, Haas M, Hestbaek L, Adams A, Bronfort G. Manual examination of the spine: a systematic critical literature review of reproducibility. J Manipulative Physiol Ther. 2006 Jul-Aug;29(6):475-85, 485.e1-10. doi: 10.1016/j.jmpt.2006.06.011. PMID 16904495
- [Background] Viikari-Juntura E. Interexaminer reliability of observations in physical examinations of the neck. Phys Ther. 1987 Oct;67(10):1526-32. doi: 10.1093/ptj/67.10.1526. PMID 3659137
- [Background] Vincent-Smith B, Gibbons P. Inter-examiner and intra-examiner reliability of the standing flexion test. Man Ther. 1999 May;4(2):87-93. doi: 10.1054/math.1999.0173. PMID 10509062
- [Background] Vroomen PC, de Krom MC, Wilmink JT, Kester AD, Knottnerus JA. Diagnostic value of history and physical examination in patients suspected of lumbosacral nerve root compression. J Neurol Neurosurg Psychiatry. 2002 May;72(5):630-4. doi: 10.1136/jnnp.72.5.630. PMID 11971050
- [Background] Wainner RS, Fritz JM, Irrgang JJ, Boninger ML, Delitto A, Allison S. Reliability and diagnostic accuracy of the clinical examination and patient self-report measures for cervical radiculopathy. Spine (Phila Pa 1976). 2003 Jan 1;28(1):52-62. doi: 10.1097/00007632-200301010-00014. PMID 12544957
- [Background] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853